CLINICAL TRIAL: NCT05248880
Title: A Phase 3 Multicenter Study to Evaluate the Safety and Efficacy of AGN-151586 for the Treatment of Glabellar Lines in Toxin-Naïve Subjects
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Intramuscular AGN-151586 Injection in Toxin-Naïve Adult Participants With Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M21-508
Record Dates: First submitted 2022-02-14; First posted 2022-02-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; AGN-151586

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGN-151586 (Experimental): Participants will receive 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1. Based on meeting the retreatment criteria, the participant may also receive 1 open-label treatment of AGN-151586.
  Interventions: Drug: AGN-151586
- Placebo (Experimental): Participants will receive 5 intramuscular injections of Placebo in the glabellar complex on Day 1. Based on meeting the retreatment criteria, the participant may also receive 1 open-label treatment of AGN-151586.
  Interventions: Drug: AGN-151586; Drug: Placebo

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular Injection
Drug: Placebo — Intramuscular Injection
  Arms: Placebo

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. AGN-151586 is an investigational product being developed for the treatment of GL. The purpose of this study is to evaluate the safety and efficacy of AGN-151586 for the treatment of GL in toxin-naïve participants with moderate to severe GL.

This is a 12 week study in which eligible subjects will be enrolled into the study containing 2 treatment periods, double-blind period and open-label period. Participants are randomly assigned to receive AGN-151586 or placebo. There is 1 in a 4 chance that participants will receive placebo. Around 300 adult participants with moderate to severe GL will be enrolled in the study in approximately 15 sites.

Participants will receive either AGN-151586 or Placebo administered as 5 intramuscular injections to the glabellar complex on Day 1. Participants meeting retreatment criteria may receive an open-label treatment of AGN-151586 during the study.

Participants will attend regular visits during the study at a study site. The effect of the treatment will be checked by medical assessments, blood tests, telephone calls, questionnaires and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to accurately assess their facial lines without the use of eyeglasses (contact lens use is acceptable).
* Participant must have moderate or severe Glabellar Lines at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale (FWS) at Screening and Baseline Day 1 visit.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Participants must not have a history of any use of botulinum neurotoxin of any serotype for any indication (including any investigational botulinum neurotoxin product).
* Presence or history of any medical condition that may place the participant at increased risk following exposure to AGN-151586 or interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the treatment injection sites
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart
  * Any eyebrow or eyelid ptosis at screening or Baseline Day 1 visit as determined by the investigator
* History of known immunization to any botulinum neurotoxin serotype.
* Tattoos, jewelry, or clothing which obscure the glabellar area and cannot be removed.
* Anticipated need for surgery or overnight hospitalization during the study.
* History of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., rhinoplasty, facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* History of periorbital, mid-facial, or upper-facial treatment with semi permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Female subject who is pregnant or breastfeeding, and is considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
* Participant who has been treated with any investigational drug within 30 days of the drug prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* Anticipated need for treatment with botulinum neurotoxin of any serotype for any reason during the study (other than study drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with ≥ 2-grade improvement from baseline on the Facial Wrinkle Scale (FWS) according to both investigator and participant assessments (composite) of Glabellar Lines (GL) severity at maximum frown | Day 7
  The investigator and participant assessments of GL severity at maximum frown using a 4-grade scale (0 to 3) where 0=none and 3=severe.
Number of Participants with Adverse Events | Up to 12 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.
Change from baseline in Vital Sign Measurements | Up to 12 Weeks
  Percentage of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change from baseline in ECG parameters | Up to 12 Weeks
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Change from baseline in laboratory evaluations | Up to 12 Weeks
  Percentage of participants with abnormal clinical laboratory values like hematology and chemistry will be assessed.
Presence of binding and neutralizing antidrug antibodies | Up to 12 Weeks
  Blood samples for immunogenicity testing will be collected from all participants treated with AGN-151586 at predetermined timepoints. Collected samples will be processed to yield serum for detection of binding and neutralizing antibodies to AGN-151586.

SECONDARY OUTCOMES:
Percentage of participants with ≥ 2-grade improvement from baseline on the FWS according to investigator assessment of GL severity at maximum frown over the double-blind period | Up to 6 Weeks
  The investigator assessment of GL severity at maximum frown using a 4-grade scale (0 to 3) where 0=none and 3=severe.
Percentage of participants with ≥ 2-grade improvement from baseline on the FWS according to participant assessment of GL severity at maximum frown over the double-blind period | Up to 6 Weeks
  The investigator assessment of GL severity at maximum frown using a 4-grade scale (0 to 3) where 0=none and 3=severe.
Percentage of participants with achievement of Mostly Satisfied or Very Satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Item 5 (overall satisfaction) for GL | Day 7
  The Facial Line Satisfaction Questionnaire assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the subject perspective.
Percentage of participants with achievement of Mostly Satisfied or Very Satisfied on the FLSQ Item 5 (overall satisfaction) for GL | Hour 24
  The Facial Line Satisfaction Questionnaire assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the subject perspective.
Percentage of participants with achievement of Mostly Satisfied or Very Satisfied on the FLSQ Item 4 (natural look) for GL | Day 7
  The Facial Line Satisfaction Questionnaire assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the subject perspective.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (17):
- United States (12):
  - Clear Dermatology & Aesthetics Center /ID# 238990, Scottsdale, Arizona
  - Steve Yoelin MD Medical Assoc. Inc /ID# 243197, Newport Beach, California
  - Marcus Facial Plastic Surgery /ID# 241703, Redondo Beach, California
  - DMR Research PLLC /ID# 239061, Westport, Connecticut
  - Kavali Plastic Surgery /ID# 244808, Atlanta, Georgia
  - Delricht Research - 10154 Jefferson /ID# 244890, Baton Rouge, Louisiana
  - Maryland Dermatology Laser, Skin, & Vein Institute /ID# 239067, Hunt Valley, Maryland
  - Wilmington Dermatology Center /ID# 233935, Wilmington, North Carolina
  - Clinical Research Center of the Carolinas /ID# 239064, Charleston, South Carolina
  - Austin Institute for Clinical Research /ID# 238989, Pflugerville, Texas
  - Kalo Clinical Research /ID# 247279, West Valley City, Utah
  - SkinDC /ID# 238988, Arlington, Virginia
- Canada (5):
  - YVR Aesthetics Training & Study Centre /ID# 241858, Vancouver, British Columbia
  - Pacific Derm /ID# 239654, Vancouver, British Columbia
  - Dr Melinda Gooderham Medicine Profession /ID# 239657, Cobourg, Ontario
  - The Centre for Clinical Trials /ID# 245873, Oakville, Ontario
  - Clinique D /ID# 239653, Laval, Quebec

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/